CLINICAL TRIAL: NCT05290259
Title: Evaluation of the Ballroom Basics for Balance Program
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0263; A176000 (Other: UW Madison); Protocol Version 3/7/2022 (Other: UW Madison)
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Balance; Gait
Keywords: ballroom dance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ballroom Basics for Balance Program: The Ballroom Basics for Balance program is a 12-week physical activity program which uses dance to focus on balance for community dwelling adults.
  Interventions: Other: Ballroom Dance

INTERVENTIONS:
Other: Ballroom Dance — The Ballroom Basics for Balance Program is a dance focused exercise program developed by a Physical Therapist in the Madison area.

SUMMARY:
The objective of this study is to evaluate the effectiveness of the 12-week Ballroom Basics for Balance (BB4B). 20 older adults in the Madison, Wisconsin area who self-select into the Ballroom Basics for Balance Program will be on study for the 12 week intervention plus pre- and post-intervention tests within 10 days for program start and completion.

DETAILED DESCRIPTION:
The primary aim is to examine how balance is impacted by participation in this program.

The secondary aims are to examine how the program impacts metrics of gait, fall frequency, occupational performance, functional cognition and functional gait. The investigators hypothesize that participation in this program will lead to significant within-subject changes from pre to post-test in both our primary and secondary outcomes.

* Hypothesis 1: Balance, as measured by the MiniBESTest, will improve (score will increase) from baseline to posttest for individuals who participate in the 12-week BB4B program.
* Hypothesis 2: Overground gait speed will increase, time spent in double support will decrease and step extremity ratio will increase from baseline to posttest.
* Hypothesis 3: Measures of occupational performance, functional cognition and functional gait will significantly improve from baseline to posttest. Fall frequency will improve non-significantly due to the limited number of participants in the study

ELIGIBILITY:
Inclusion Criteria:

* Individuals enrolled in the BB4B program
* Volunteered for the research study
* Scored a 25 or higher on the Montreal Cognitive Assessment (MoCA), indicating that no cognitive impairment is present.
* English speaking

Exclusion Criteria:

* children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults in the Madison area who self-select into the Ballroom Basics for Balance Program
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Change in Activities-Specific Balance Confidence Scale (ABC) | baseline, posttest (up to 14 weeks)
  16-item survey of how confident one is with balance, scored as a percentage between 0-100 where higher percentage indicates increased confidence in balance.
Change in Falls Efficacy Scale (FES) | baseline, posttest (up to 14 weeks)
  10-item survey that measures confidence in one's own ability to complete daily activities without falling on a scale of 1-10 where lowers scores indicate more extreme confidence.
Change in the Mini-BESTest Score | baseline, posttest (up to 14 weeks)
  The mini-BESTest will be used to assess balance. This 14-item, clinical battery is used to assess balance in four component areas (anticipatory transitions, postural response, sensory orientation and dynamic gait) and provides a single number summary of balance performance (total possible range of scores 0-30), higher scores indicate better balance.

SECONDARY OUTCOMES:
Change in Spatiotemporal measures of gait: Gait Speed | baseline, posttest (up to 14 weeks)
  The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support.
  Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem (one foot directly in front of the other (heel to toe)) and dual task (naming items in a specified category) gait. Each participant will complete up to 10 trials for each condition.
Change in Spatiotemporal measures of gait: percent of cycle in double support | baseline, posttest (up to 14 weeks)
  The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support.
  Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem (one foot directly in front of the other (heel to toe)) and dual task (naming items in a specified category) gait. Each participant will complete up to 10 trials for each condition.
Change in Spatiotemporal measures of gait: Base of Support measured as horizontal stride width | baseline, posttest (up to 14 weeks)
  The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support.
  Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem (one foot directly in front of the other (heel to toe)) and dual task (naming items in a specified category) gait. Each participant will complete up to 10 trials for each condition.
Change in Spatiotemporal measures of gait: Stride Length | baseline, posttest (up to 14 weeks)
  The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support.
  Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem (one foot directly in front of the other (heel to toe)) and dual task (naming items in a specified category) gait. Each participant will complete up to 10 trials for each condition.
Change in Spatiotemporal measures of gait: Cadence in steps per minute | baseline, posttest (up to 14 weeks)
  The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support.
  Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem (one foot directly in front of the other (heel to toe)) and dual task (naming items in a specified category) gait. Each participant will complete up to 10 trials for each condition.
Change in Fall Frequency | baseline, posttest (up to 14 weeks)
  At baseline and posttest, participants will be asked to estimate their fall frequency (none, 1 time, 2-10 times, weekly, daily) in the last 2 weeks, 1 month, and 6 months.
Change in Canadian Occupational Performance Measure (COPM): Performance Score | baseline, posttest (up to 14 weeks)
  Total possible range of scores from 1-10 where higher scores indicate higher performance.
Change in Canadian Occupational Performance Measure (COPM): Satisfaction Score | baseline, posttest (up to 14 weeks)
  Total possible range of scores from 1-10 where higher scores indicate higher satisfaction.

OTHER OUTCOMES:
Change in Menu Task Score | baseline, posttest (up to 14 weeks)
  The Menu Task is a performance based screening tool used to examine functional cognition. Total scores will range between 0-12 where higher scores indicate increased functional cognition.
Change in Functional Gait measured by Performance Assessment of Self-Care Skills (PASS) | baseline, posttest (up to 14 weeks)
  Specific components of the the PASS assessment will be administered to examine changes in performance of activities of daily living. The PASS consists of 26 activities of daily living and is designed to allow for a client-centered, performance-based means of objectively assessing occupation-based interventions. A modified version of the shopping component of the PASS assessment will be performed in an instrumented environment (SMIL kitchen) to allow for quantification of kinetic and kinematic measures relative to the performance of these tasks.
  Scores will range from 0-3 on individual metrics where higher numbers indicate increased independence, safety, and adequacy. Spatiotemporal gait measures will be used for quantitative scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Pickett, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Sensory Motor Integration Lab, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Pickett will be responsible for deciding when/to whom to disseminate coded data, and will work with other researchers if necessary to confirm that they have proper IRB approval/etc., as necessary. Required UW-Madison IRB approval would be obtained prior to the release of any data.
Supporting Information: Study Protocol, SAP, ICF